CLINICAL TRIAL: NCT03461237
Title: Second Hip Fracture Evaluation in Chinese Elderly Patients Using Quantitative Computed Tomography
Brief Title: Chinese Second Hip Fracture Evaluation
Acronym: CSHFE
Status: Recruiting | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, xiaoguang Cheng, Chairman, Department of Radiology, Beijing Jishuitan Hospital
Other Study IDs: JST2016CSHFE
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Osteoporosis
Keywords: Second Hip Fracture; Quantitative Computed Tomography; Bone structure; Muscle
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
1. To Compare overall rates of second hip fractures in both genders,
2. To determine the effect of hip fracture on proximal femoral volumetric bone mineral density (vBMD), bone structure and muscle by quantitative computed tomography(QCT),
3. To evaluate the contribution of QCT-image analysis to the prediction of the second hip fracture risk.
4. To identify the differences between femoral neck fracture and trochanter fracture following hip fracture

DETAILED DESCRIPTION:
Osteoporotic hip fracture is a great harm among elderly people, for whom disability and death often occurs. Furthermore, sustaining an osteoporotic hip fracture increases the risk of a subsequent fracture. However, the risk factors of subsequent hip fractures are less studied and the proximal femur bone structure and muscle changes following first hip fracture are little known.

Therefore, we propose to conduct an observational and perspective study to assess the effect of hip fracture on proximal femoral bone and muscle using quantitative computed tomography (QCT), as well as to evaluate the contribution of QCT-image analysis to the prediction of the second hip fracture risk. As hip fractures are divided into two major anatomic based types in clinical: femoral neck fractures (intracapsular) and trochanter fractures (extracapsular), the fundamental objective also includes identifying bone and muscle differences in a union activity between the two type fractures. Compared with duel-energy x-ray absorptiometry (DXA), QCT offers the advantage of selective measurement of the metabolically active and structurally important trabecular bone in the proximal femoral. Volumetric BMD and structure of proximal femoral and muscle around hip will be measured with QCT. The CT scanner will be the clinical CT scanner of the local participated center. Quality control and monitoring will be conducted by Beijing Jishuitan hospital, as well as the centralised image interpretation.

ELIGIBILITY:
Inclusion Criteria:

* a:Osteoporotic patients b:Osteoporotic hip fracture patients (femoral neck fracture and femoral trochanteric fracture) c: Be willing to and be able to join in the study and sighed the informed consent

Exclusion Criteria:

* a:Under 47years old b:Non-surgical repair of hip fracture c:Pathologic fracture d:Violence-related trauma e:Bilateral hip implants or have hip replacement on the non-fractured side

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cohort-based study. 3000 participants (including 1800 females and 1200 males) who (>47 years old) have recently suffered single hip fracture will be recruited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Hip re-fracture | 3 years
  The incidence and location of second hip fracture
all cause death | 2 year
  all cause death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoguang Cheng, MD, Principal Investigator — department of radiology, Beijing Jishuitan Hospital
Locations (1):
- Beijing ji shui tan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma Y, Ge Y, Guo Z, Su Y, Wang C, Wang Q, Wang L, Cheng X, Yang M, Yan D. Hip structural analysis parameters are not associated with the risk of postmenopausal female second hip fracture: a retrospective study. BMC Musculoskelet Disord. 2025 Mar 10;26(1):233. doi: 10.1186/s12891-025-08368-7. PMID 40065296